CLINICAL TRIAL: NCT06461377
Title: The Ameliorative Effects of GLP-1RA on Diabetic Cardiac Autonomatic Neuropathy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-SR-611
Record Dates: First submitted 2024-03-01; First posted 2024-06-17 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Type 2 Diabetes; Diabetes With Diabetic Autonomic Neuropathy (Diagnosis)
Keywords: T2DM，DCAN，HRV, CART，insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Disease | interventions — semaglutide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): In the control group, no other intervention was used except the basic drugs for diabetes treatment
- GLP-1RA intervention group (Experimental): Subcutaneous injection of semaglutide 0.5-1mg （dosage depends on individual body weight）once a week (not off-label use)，lasting 12 weeks
  Interventions: Drug: Glucagon-like peptide-1 receptor agonist：Semaglutide

INTERVENTIONS:
Drug: Glucagon-like peptide-1 receptor agonist：Semaglutide — The GLP-1RA intervention group was given subcutaneous injection of GLP-1RA for 3 months, while the control group was not given GLP-1RA intervention
  Other Names: Semaglutide
  Arms: GLP-1RA intervention group

SUMMARY:
Diabetic cardiac autonomic neuropathy (DCAN) is a common chronic complication that reduces survival in patients with diabetes. Epidemiological surveys have shown that the prevalence of DCAN is 25-75% in people with type 2 diabetes. The onset of DCAN is insidious and easy to be ignored in the early stage. With the progression of the disease, the following clinical symptoms gradually appear, including reduced heart rate variability, exercise intolerance, resting tachycardia, orthostatic hypotension, painless myocardial infarction and even sudden death, which seriously endanger the life and health of type 2 diabetes patients. Existing literature has shown that glucagon-like peptide-1 receptor agonist (GLP-1RA) can improve diabetic peripheral neuropathy and diabetic cognitive dysfunction, but there are few studies on improving diabetic autonomic neuropathy. Insulin resistance is an important risk factor for DCAN. Patients with type 2 diabetes are characterized by insulin resistance, and GLP-1RA is recognized as a drug to improve insulin resistance and control blood sugar in patients with diabetes. In this study, GLP-1RA was used to intervene patients with type 2 diabetes, and the changes in blood sugar control and insulin resistance status of patients were followed up. Special attention was paid to the improvement of autonomic neuropathy in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-70 years
2. Patients with T2DM who meet the diagnostic guidelines
3. The patient signed the relevant informed consent form
4. Being overweight or obese

Exclusion Criteria:

1. <18 years old
2. Pregnant or lactating women
3. Acute and chronic pancreatitis
4. Recent acute complications of diabetes
5. Arrhythmia or taking drugs that affect heart rate
6. Thyroid disease
7. Severe organ dysfunction
8. Denial of informed consen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
heart rate variability（HRV） | baseline and 12 weeks later
  All participants were given ambulatory electrocardiogram.The time domain analysis and frequency domain analysis of heart rate variability are included in the holter ECG report.

SECONDARY OUTCOMES:
E/I difference | basline and 12 weeks later
  Take an average of 6 deep breaths per minute, record the difference between the maximum heart rate and the minimum heart rate during deep breathing
30/15 ratio | basline and 12 weeks later
  The heart rate in lying position was measured, and the R-R interval in more than 30 beats was measured after standing, and the ratio between the longest R-R interval in the 25-35 beats and the shortest R-R interval in the 10-15 beats after standing was calculated
Valsalva action | basline and 12 weeks later
  After deep inhalation, hold your breath as much as possible, and then blow air into the modified sphygmomanometer to keep the pressure of the sphygmomanometer at 40mmHg, continue for 10-15s, and then relax for 1 minute, a total of 3 minutes. At the same time, ECG was recorded to record the ratio of maximum heart rate to minimum heart rate
the difference between lying and Orthostatic blood pressure | basline and 12 weeks later
  Blood pressure was measured in the supine position. The patient was asked to stand immediately, and blood pressure was measured at the first and fifth minutes
grip strength tests | basline and 12 weeks later
  First, the basic blood pressure and the maximum grip strength were measured, and the blood pressure was measured after 5 minutes of continuous hard clenching with the grip apparatus (the force used was 30% of the maximum grip strength measured), and the blood pressure difference was calculated
BMI | basline and 12 weeks later
  It is calculated by dividing a person's weight in kg by their height in meters squared
FBG | basline and 12 weeks later
  Fasting glucose
Fins | basline and 12 weeks later
  Fasting insulin
Fc-peptide | basline and 12 weeks later
  Fasting c-peptide
HOMA-IR | basline and 12 weeks later
  calculated by HOMA Calculator v2.2.3
HbA1c | basline and 12 weeks later
  Reflect the average blood sugar of 3 months
Total cholesterol | basline and 12 weeks later
  one of serum biochemical index
triglyceride | basline and 12 weeks later
  one of serum biochemical index
HDL | basline and 12 weeks later
  high-density lipoprotein，one of serum biochemical index
LDL | basline and 12 weeks later
  low density lipoprotein，one of serum biochemical index
UA | basline and 12 weeks later
  Uric Acid，one of serum biochemical index
creatinine | basline and 12 weeks later
  one of serum biochemical index
eGFR | basline and 12 weeks later
  Estimated glomerular filtration rate，one of serum biochemical index
Urinary trace albumin/urinary creatinine | basline and 12 weeks later
  urine protein test urine protein urine protein test

CONTACTS AND LOCATIONS:
Overall Officials: jianbo Li, MD/PhD, Principal Investigator — First Affiliated Hospital，Nanjing Medical University，China
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Maser RE, Lenhard MJ. Cardiovascular autonomic neuropathy due to diabetes mellitus: clinical manifestations, consequences, and treatment. J Clin Endocrinol Metab. 2005 Oct;90(10):5896-903. doi: 10.1210/jc.2005-0754. Epub 2005 Jul 12. PMID 16014401
- [Background] Balcioglu AS, Muderrisoglu H. Diabetes and cardiac autonomic neuropathy: Clinical manifestations, cardiovascular consequences, diagnosis and treatment. World J Diabetes. 2015 Feb 15;6(1):80-91. doi: 10.4239/wjd.v6.i1.80. PMID 25685280
- [Background] Vinik AI, Maser RE, Mitchell BD, Freeman R. Diabetic autonomic neuropathy. Diabetes Care. 2003 May;26(5):1553-79. doi: 10.2337/diacare.26.5.1553. PMID 12716821
- [Background] Goh JK, Koh L. Evaluating treatment options for cardiovascular autonomic neuropathy in patients with diabetes mellitus: a systematic review. Diabetol Int. 2023 Apr 25;14(3):224-242. doi: 10.1007/s13340-023-00629-x. eCollection 2023 Jul. PMID 37397902
- [Background] Kaze AD, Yuyun MF, Fonarow GC, Echouffo-Tcheugui JB. Cardiac autonomic dysfunction and risk of incident stroke among adults with type 2 diabetes. Eur Stroke J. 2023 Mar;8(1):275-282. doi: 10.1177/23969873221127108. Epub 2022 Nov 1. PMID 37021204
- [Background] Williams SM, Eleftheriadou A, Alam U, Cuthbertson DJ, Wilding JPH. Cardiac Autonomic Neuropathy in Obesity, the Metabolic Syndrome and Prediabetes: A Narrative Review. Diabetes Ther. 2019 Dec;10(6):1995-2021. doi: 10.1007/s13300-019-00693-0. Epub 2019 Sep 24. PMID 31552598
- [Background] Dimitropoulos G, Tahrani AA, Stevens MJ. Cardiac autonomic neuropathy in patients with diabetes mellitus. World J Diabetes. 2014 Feb 15;5(1):17-39. doi: 10.4239/wjd.v5.i1.17. PMID 24567799
- [Background] Wink J, van Delft R, Notenboom RGE, Wouters PF, DeRuiter MC, Plevier JWM, Jongbloed MRM. Human adult cardiac autonomic innervation: Controversies in anatomical knowledge and relevance for cardiac neuromodulation. Auton Neurosci. 2020 Sep;227:102674. doi: 10.1016/j.autneu.2020.102674. Epub 2020 May 16. PMID 32497872
- [Background] Kapa S, DeSimone CV, Asirvatham SJ. Innervation of the heart: An invisible grid within a black box. Trends Cardiovasc Med. 2016 Apr;26(3):245-57. doi: 10.1016/j.tcm.2015.07.001. Epub 2015 Jul 9. PMID 26254961
- [Background] Aksu T, Gupta D, Pauza DH. Anatomy and Physiology of Intrinsic Cardiac Autonomic Nervous System: Da Vinci Anatomy Card #2. JACC Case Rep. 2021 Apr 21;3(4):625-629. doi: 10.1016/j.jaccas.2021.02.018. eCollection 2021 Apr. PMID 34317590
- [Background] Kikel-Coury NL, Brandt JP, Correia IA, O'Dea MR, DeSantis DF, Sterling F, Vaughan K, Ozcebe G, Zorlutuna P, Smith CJ. Identification of astroglia-like cardiac nexus glia that are critical regulators of cardiac development and function. PLoS Biol. 2021 Nov 18;19(11):e3001444. doi: 10.1371/journal.pbio.3001444. eCollection 2021 Nov. PMID 34793438
- [Background] Jorgensen JR, Thompson L, Fjord-Larsen L, Krabbe C, Torp M, Kalkkinen N, Hansen C, Wahlberg L. Characterization of Meteorin--an evolutionary conserved neurotrophic factor. J Mol Neurosci. 2009 Sep;39(1-2):104-16. doi: 10.1007/s12031-009-9189-4. Epub 2009 Mar 4. PMID 19259827
- [Background] Lee HS, Han J, Lee SH, Park JA, Kim KW. Meteorin promotes the formation of GFAP-positive glia via activation of the Jak-STAT3 pathway. J Cell Sci. 2010 Jun 1;123(Pt 11):1959-68. doi: 10.1242/jcs.063784. Epub 2010 May 11. PMID 20460434
- [Background] Mehta K, Behl T, Kumar A, Uddin MS, Zengin G, Arora S. Deciphering the Neuroprotective Role of Glucagon-like Peptide-1 Agonists in Diabetic Neuropathy: Current Perspective and Future Directions. Curr Protein Pept Sci. 2021;22(1):4-18. doi: 10.2174/1389203721999201208195901. PMID 33292149
- [Background] Takaku S, Tsukamoto M, Niimi N, Yako H, Sango K. Exendin-4 Promotes Schwann Cell Survival/Migration and Myelination In Vitro. Int J Mol Sci. 2021 Mar 15;22(6):2971. doi: 10.3390/ijms22062971. PMID 33804063